CLINICAL TRIAL: NCT03071315
Title: Economic Evaluation Comparing Center-based Compulsory Drug Treatment With Community-based Methadone Maintenance Treatment in Hai Phong City, Vietnam
Brief Title: Economic Evaluation Comparing CCT With MMT in Hai Phong City, Vietnam
Status: Completed | Type: Observational
Sponsor: The University of New South Wales (Other)
Collaborators: The Atlantic Philanthropies (Other); FHI 360 (Other); Hanoi Medical University (Other); University of Adelaide (Other)
Responsible Party: Principal Investigator, Alison Ritter, Professor, The University of New South Wales
Other Study IDs: HC12259
Record Dates: First submitted 2017-02-28; First posted 2017-03-06 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Heroin Dependence
Keywords: Economic evaluation; Heroin dependence; Compulsory treatment; Methadone treatment; Vietnam; East and Southeast Asia; Cost-effectiveness
MeSH Terms: conditions — Heroin Dependence | interventions — 2-methylcyclopentadienyl manganese tricarbonyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCT participants: Center-based compulsory treatment (CCT) participants who were placed into compulsory treatment centers for two years for a range of punitive treatment such as education, moral teaching, labor work. Very basic health care is provided in the CCT centers.
  Interventions: Other: CCT
- MMT participants: Methadone maintenance treatment (MMT) participants who have been receiving MMT treatment. In Hai Phong City, during the period of this study, voluntary MMT was provided in the community free for people who were assessed as dependent on heroin.
  Interventions: Other: MMT

INTERVENTIONS:
Other: CCT — CCT focuses on behavioral approach, mainly punitive punishment measures.
  Groups: CCT participants
Other: MMT — MMT is a combination of pharmaceutical and behavioral intervention.
  Groups: MMT participants

SUMMARY:
The study compared the effectiveness and cost-effectiveness of two dominant heroin dependence treatment approaches: center-based compulsory rehabilitation (CCT) and community-based voluntary methadone treatment (MMT) in Hai Phong City, Vietnam. The design was a combined retrospective and prospective, non-randomized cohort over three years (with data at five time-points). The study was conducted between 2012 and 2015, involving 208 CCT participants and 384 MMT participants with heroin dependence.

DETAILED DESCRIPTION:
The study compared the effectiveness and cost-effectiveness of two dominant heroin dependence treatment approaches: center-based compulsory rehabilitation (CCT) and community-based voluntary methadone treatment (MMT) in Hai Phong City, Vietnam. CCT centers are institutions in which people who use drugs are confined for two years. MMT has been internationally recognized as an efficacious treatment for heroin dependence and was introduced in Vietnam in 2008.

The design was combined retrospective and prospective, non-randomized cohort over three years (with data at five time-points). The study was conducted between 2012 and 2014, involving 208 CCT participants (of which 80% were followed up) and 384 MMT participants (of which 78% were followed up) with heroin dependence. The five time-points were: baseline, two years after treatment commencement, then three months, six months and 12 months after the initial two years. The study combined primary data and secondary data to assess the effectiveness of the two treatment modalities. The economic component measured the costs of the two treatment modalities to compare cost-effectiveness outcomes.

The study had two primary outcomes: self-reported heroin abstinence (confirmed by urine drug screening) and self-reported drug-free days (DFDs). DFDs was reported in two different time-frames. DFDs in the preceding 30 days was used for effectiveness comparison and DFDs over three years was used for the cost-effectiveness comparison. The study has four secondary outcomes: illegal behaviors, overdose, blood-borne virus (BBV) risk behaviors, and monthly drug spending).

Mixed effects regression models were used to analyze the effectiveness data and non-parametric bootstrapping methods were used to estimate cost-effectiveness. The time-frame for the cost-effectiveness analysis was three years.

ELIGIBILITY:
Inclusion Criteria (for CCT Participants):

* 18 years of age and older
* Heroin dependent
* CCT-released participants who were rehabilitated in the CCT centers under the compulsory track.
* CCT-released participants who received the recruitment letter sent by CCT centers' staff and who could provide either the recruitment letter or a certificate of CCT treatment completion at the time of first contact with a researcher as a proof that they were newly CCT-released participants.
* Consented voluntarily to participate in the study, as assessed and determined by the researcher providing the informed consent documentation.

Exclusion Criteria (for CCT Participants):

* Younger than 18 years old
* Severe cognitive or mental impairment
* Unable to grant consent for this research study
* Non-dependent use of heroin.

Inclusion Criteria (for MMT Participants):

* 18 years of age and older
* Heroin dependence, measured by self-reported daily use of heroin during 3 months prior to index treatment, a proxy to measure heroin dependence
* Participated in MMT treatment in Hai Phong City from 2008-2009
* Consented voluntarily to participate in this research, as assessed and determined by the researcher providing the informed consent documentation.

Exclusion Criteria (for MMT Participants):

* Younger than 18 years old
* Severe cognitive or mental impairment
* Unable to grant consent for this research study
* Non-dependent use of heroin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CCT Participants: Participants who were placed in three CCT centers in Hai Phong City for 2 years (2011-2013) and agreed to voluntarily participate in this study (from July 2013: 12 months community follow-up).
  MMT Participants: Participants who have participated in a previous cohort study (two-years:2009-2012) and agreed to voluntarily participate in this study (from 2013: an addition of 12 months)
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2013-01-20 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Heroin abstinence | Preceding 3 months and 30 days
  Free from heroin use (self-reported), confirmed by urine drug screening on interview day.

SECONDARY OUTCOMES:
Drug-free days | Preceding 3 months and 30 days
  Days without use of any illicit drugs (self-report)
Drug-use related illegal behaviors | Preceding 3 months and 30 days
  Drug-use related illegal behaviors
Drug-use related blood-borne virus (BBV) risk behaviors | Preceding 3 months and 30 days
  Drug-use related blood-borne virus (BBV) risk behaviors
Overdose incidents | Preceding 3 months and 30 days
  Overdose incidents
Monthly drug spending | Preceding 3 months and 30 days
  Monthly drug spending

CONTACTS AND LOCATIONS:
Overall Officials: Alison Ritter, PhD, Principal Investigator — The University of New South Wales
Locations (1):
- Study site in Vietnam, Haiphong, Hai Phong, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vuong T, Ritter A, Shanahan M, Ali R, Nguyen N, Pham K, Vuong TTA, Le GM. Outcomes of compulsory detention compared to community-based voluntary methadone maintenance treatment in Vietnam. J Subst Abuse Treat. 2018 Apr;87:9-15. doi: 10.1016/j.jsat.2018.01.011. Epub 2018 Jan 16. PMID 29471930